CLINICAL TRIAL: NCT00170937
Title: A 16 Week Study to Evaluate the Effect on Insulin Sensitivity of Valsartan and Hydrochlorothiazide Combined and Alone, in Patients With Metabolic Syndrome
Brief Title: A 16 Week Study to Evaluate the Effect on Insulin Sensitivity of Valsartan (320 mg) and Hydrochlorothiazide (25 mg) Combined and Alone, in Patients With Metabolic Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CVAL489A2426
Record Dates: First submitted 2005-09-10; First posted 2005-09-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: METABOLIC SYNDROME; HYPERTENSION; PRE-HYPERTENSION
Keywords: METABOLIC SYNDROME, VALSARTAN, HYDROCHLOROTHIAZIDE, HYPERTENSION,
MeSH Terms: conditions — Metabolic Syndrome; Hypertension; Prehypertension | interventions — Valsartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: valsartan plus hydrochlorothiazide

SUMMARY:
The metabolic syndrome is a classification for patients with a constellation of risk factors which may include abdominal obesity, hypertension, elevated blood lipids and sugar. Three or more of these factors together constitute the metabolic syndrome and place these patients at a greater risk for the development of diabetes and cardiovascular diseases. The purpose of this study is to determine whether two common drugs to lower blood pressure, whether used separately or in combination, have different effects on blood sugar levels in patients diagnosed with the metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Waist circumference: males > 40", females > 35 "
* MSSBP ≥ 130 mmHg but ≤ 160 mmHg and a MSDBP ≥ 85 mmHg but ≤ 100 mmHg
* At least one of the following criteria: - Fasting plasma glucose between 5.9 and 6.9 mmol/L; - Serum triglycerides > 150 mg/dL; - LDL Cholesterol: - < 40 mg/dL males; - < 50 mg/dL females

Exclusion Criteria:

* MSSBP> 180 mmHg or MSDBP > 110 mmHg
* Inability to discontinue all prior antihypertensives for a period of 4 weeks.
* History of diabetes
* History of stroke, transient ischemic attack or myocardial infarction.
* Significant weight change > 10 lbs during screening period
* Patients taking a diuretic for 3 months prior to screening.

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 507
Dates: Start 2004-11; Primary Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity after 16 weeks

SECONDARY OUTCOMES:
Change from baseline in markers of inflammation and thrombosis after 16 weeks
Change from baseline in fasting plasma glucose and fasting insulin after 16 weeks
Change from baseline in lipid profile after 16 weeks
Change from baseline in a measurement of beta cell function after 16 weeks
Adverse events, serious adverse events, laboratory values, physical examinations, and vital signs for up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States

REFERENCES:
- [Result] Zappe DH, Sowers JR, Hsueh WA, Haffner SM, Deedwania PC, Fonseca VA, Keeling L, Sica DA. Metabolic and antihypertensive effects of combined angiotensin receptor blocker and diuretic therapy in prediabetic hypertensive patients with the cardiometabolic syndrome. J Clin Hypertens (Greenwich). 2008 Dec;10(12):894-903. doi: 10.1111/j.1751-7176.2008.00054.x. PMID 19120715